CLINICAL TRIAL: NCT07024342
Title: Optimizing Prosthetic Prescription to Mitigate the Effects of Perspiration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Glenn K. Klute, PhD, Research Career Scientist / Affiliate Professor, VA Puget Sound Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1588234
Record Dates: First submitted 2022-06-02; First posted 2025-06-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Amputation; Prosthesis User
Keywords: Lower limb prosthesis; perspiration; adherence

STUDY DESIGN:
Intervention Model Description: A between-subjects, repeated measures experiment will be conducted with individuals with unilateral transtibial limb loss (n=180) who are successful ambulators and have issues with perspiration by self-report. Baseline measurements will be obtained at the time of enrollment while participants are wearing their as-prescribed liner. After wearing the randomly assigned study intervention for two weeks, measurements will be repeated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Liner perforated with very small diameter holes (Experimental): Subjects will wear their prosthesis in their home, work, and community environments while they will participate in their usual activities for two weeks.
  Interventions: Device: Liner perforated with very small diameter holes; Device: As-prescribed liner
- Liner perforated with somewhat larger diameter holes (Experimental): Subjects will wear their prosthesis in their home, work, and community environments while they will participate in their usual activities for two weeks.
  Interventions: Device: Liner perforated with somewhat larger diameter holes; Device: As-prescribed liner
- Liner-liner (Experimental): Subjects will wear their prosthesis in their home, work, and community environments while they will participate in their usual activities for two weeks.
  Interventions: Device: Liner-liner; Device: As-prescribed liner

INTERVENTIONS:
Device: Liner perforated with very small diameter holes — A commercially available, elastomeric liner perforated with very small holes (approximately 0.3 mm diameter) to allow perspiration to drain. This liner is worn between the skin and the participant's prosthetic socket.
  Other Names: SoftSkin Air S30; Uniprox, Zeulenroda-Triebes, GER
  Arms: Liner perforated with very small diameter holes
Device: Liner perforated with somewhat larger diameter holes — A commercially available, elastomeric liner perforated with somewhat larger holes (approximately 1.5 mm diameter) to allow perspiration to drain. This liner is worn between the skin and the participant's prosthetic socket.
  Other Names: Silcare Breathe Cushion Liner; Endolite, Miamisburg, OH, USA
  Arms: Liner perforated with somewhat larger diameter holes
Device: Liner-liner — A thin, special purpose half-ply sock which may reduce the effects of perspiration. The liner-liner is worn between the skin and the participant's as-prescribed liner.
  Other Names: Liner-liner; Knit-Rite, Kansas City, KS, USA
  Arms: Liner-liner
Device: As-prescribed liner — A commercially available, elastomeric liner with no perforations. This liner is worn between the skin and the participant's prosthetic socket.
  Other Names: Alpha Classic or Alpha Hybrid; WillowWood; Mt. Sterling, OH, USA

SUMMARY:
The specific aim of this research is to compare three clinically available liners, each intended to address problems of residual limb perspiration, with the as-prescribed liner of lower limb prosthesis user and determine their effect on stability, suspension, and comfort.

DETAILED DESCRIPTION:
The objective of the proposed research is to provide the individual with a below-knee amputation a prosthesis that best addresses problems of perspiration and its accumulation inside the prosthesis. A concern of every individual with a lower limb prosthesis is keeping their residual limb healthy and injury free. Naturally occurring perspiration, induced by moderate to vigorous activity or hot and humid environments, leads to perspiration. While the modern prosthetic liner can be stable, secure, and comfortable when dry, the materials from which they are made trap heat and are impermeable to moisture. When perspiration accumulation is a frequent occurrence, a host of biomechanical and skin problems can arise. Clinicians have few available options to prevent perspiration accumulation inside the prosthesis.

For individuals who do have problems with residual limb perspiration, some may be able to stop their activity when it accumulates, remove their prosthesis, dry it and their residual limb, then don it again and carry on. Others, like the military service personnel, may not have such an opportunity. These individuals can be prescribed a perforated liner through which perspiration can drain, or a thin, special purpose half-ply sock worn between the skin and liner, which can reduce the lubricating effects of perspiration. Current commercially-available perforated liners come with two different sized holes: one with small holes the size of a pinprick, and one with somewhat larger holes the size of a pinhead. There is little evidence available to suggest which of the three approaches is best.

The aim of the proposed research is to compare these three clinically-available options and determine which is best at addressing the problem of perspiration accumulation inside the prosthesis. To achieve this aim, we propose to recruit 180 individuals with below-knee amputations to participate in a human subject experiment. Upon enrollment, we will administer a survey to measure the stability, suspension, and comfort of their socket. Subjects will then receive one of three study-provided liners: (1) a liner-liner, (2) a liner perforated with very small diameter holes, or (3) a liner perforated with somewhat larger diameter holes. After subjects have worn the study-provided liner for two weeks, we will administer the survey again. The results of this research will identify which of the three clinically-available options is best at addressing the problem of perspiration accumulation inside the prosthesis.

More than half a million Americans live with a lower limb amputation, and a few thousand of these were on active duty when it happened. For the many individuals with a lower limb amputation who have problems with perspiration, the results of this two-year study will be of value as it will help them, and their clinicians, choose the best commercially-available solution.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation
* Been fit with a prosthesis and used it for at least six months
* Wear the prosthesis for four or more hours on average per day
* Have, or will have access to a computer, tablet, or smartphone with video conferencing ability
* Currently have problems with residual limb perspiration
* Currently wear a WillowWood Alpha Classic or Alpha Hybrid liner

Exclusion Criteria:

* Improper fit and suspension with current prosthesis and one cannot be achieved with clinical resources
* Residual limb is ulcerated
* Current skin irritation or injury on residual limb
* Osteoarthritis, injury, or pain that interferes with walking ability
* Currently incarcerated
* Pregnant
* Inadequate cognitive function or language proficiency to consent to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Difference in CLASS stability score | A baseline measurement of the CLASS stability score will be obtained upon enrollment and repeated after the subject has worn one of the study-provided liners for two weeks
  The Comprehensive Lower-limb Amputee Socket Survey (CLASS) is a self-report instrument that measures prosthesis stability, suspension, comfort, and appearance with very good internal consistency. The stability score measures how stable and balanced a person feels in their socket when they sit, stand, walk, and ascend or descend stairs.
Difference in CLASS suspension score | A baseline measurement of the CLASS suspension score will be obtained upon enrollment and repeated after the subject has worn one of the study-provided liners for two weeks
  The Comprehensive Lower-limb Amputee Socket Survey (CLASS) is a self-report instrument that measures prosthesis stability, suspension, comfort, and appearance with very good internal consistency. The suspension score measures how secure a person feels in their socket with no excessive movement when they sit, stand, walk, and ascend or descend stairs.
Difference in CLASS comfort score | A baseline measurement of the CLASS comfort score will be obtained upon enrollment and repeated after the subject has worn one of the study-provided liners for two weeks
  The Comprehensive Lower-limb Amputee Socket Survey (CLASS) is a self-report instrument that measures prosthesis stability, suspension, comfort, and appearance with very good internal consistency. The comfort score measures how comfortable a person feels in their socket when they sit, stand, walk, and ascend or descend stairs.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn K Klute, PhD, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset in machine-readable format will be created and shared for all individual participant data (IPD) that underlie results in a publication. The investigators will follow 164.514(a) of the HIPAA Privacy Rule for de-identification of IPD.
Time Frame: Within six months after publication of final study findings.
Access Criteria: Open-source data repository (e.g., PubMed Central)